CLINICAL TRIAL: NCT03027661
Title: Para-cervical Block Prior to Laparoscopic Hysterectomy as an Adjuvant Treatment to Reduce Postoperative Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-130
Record Dates: First submitted 2017-01-17; First posted 2017-01-23 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2017-01

CONDITIONS: Pain, Postoperative
Keywords: para-cervical block; laparoscopic hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Injection of 10 mL of 0.9% sodium chloride into the cervical stroma divided between 3 and 9 o'clock
  Interventions: Drug: 0.9% Sodium Chloride
- Study Group (Active Comparator): Injection of 10 mL of 0.5% bupivacaine into the cervical stroma divided between 3 and 9 o'clock.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Inject 10 mL of 0.5% bupivacaine into cervical stroma
  Other Names: Marcaine; Sensorcaine
  Arms: Study Group
Drug: 0.9% Sodium Chloride — Inject 10 mL of 0.9% NaCl into cervical stroma
  Other Names: Normal Saline
  Arms: Control Group

SUMMARY:
This is a prospective randomized controlled trial in which patients that are scheduled to undergo a laparoscopic hysterectomy would be allocated to one of two groups: Paracervical block with local anesthetic (bupivacaine 0.5%), or placebo. This would be achieved using block randomization. The intervention would be performed after the patient is under general anesthesia, prior to starting the surgery. Patients would be consented in the office or preoperative area (before receiving sedatives). As far as the intervention itself, it would consist of injecting 5 mL of 0.5% bupivacaine into the cervical stroma at 3 and 9 o'clock, which is standard technique for para-cervical block. The remainder of the procedure will then continue in a regular fashion. Alternatively, patients in the control group will be injected with 5 mL of normal saline. The surgeon would be blinded as to patient allocation. Research staff will have previously prepared the formulations (saline or bupivacaine) and have sent them to the operating room prior to beginning the procedure depending on assigned group. At the end of the case, pain will be assessed using a visual analogue scale with a range from 0 to 10 by one of the researches who will also be blinded to the group. This will be done at 30 and 60 minutes after surgical stop time. Additional pain control in the postanesthesia care unit (PACU) will be standardized to all patients.

Hypothesis:

Performing a para-cervical block with local anesthetic prior to a laparoscopic hysterectomy significantly reduces pain after the procedure

DETAILED DESCRIPTION:
Specific aims:

-Determine if infiltrating the cervical stroma with local anesthetic prior to performing a hysterectomy will reduce postoperative pain scores, and hence increase patient satisfaction.

Secondary aims:

* Determine if there is a difference in baseline pain depending on additional procedures performed, and their response to the paracervical block.
* Determine if there is a difference in response to paracervical block based on history of cesarean deliveries or uterine weight.

Background/Significance:

Hysterectomy is one of the most common surgical procedures performed in the United States, with more than 600,000 done annually. Over the last decade, there has been major changes in regards to the surgical approach utilized. With the advent of laparoscopy and robotic surgery, the rate of procedures done vaginally or abdominally has decreased significantly. One of the major drivers to this change is the demand for a faster recovery and decreased postoperative discomfort. Additionally, several adjuvant methods such as a TAP (transverse abdominal plain) block, ERAS (expedited recovery after surgery) pathway, etc. have been developed in order to minimize pain after surgery and hence increase patient satisfaction. Paracervical block is a particular technique that has been evaluated in multiple studies as a way to reduce pain after vaginal surgery. Studies have been successful in demonstrating an improvement in pain scores after these types of procedures. However, to our knowledge, there has never been follow-up to evaluate this method during the laparoscopic approach, with or without robotic assistance. The rationale of why this technique may be beneficial during a hysterectomy is that after infiltrating the cervical stroma with local anesthetic, it will diffuse towards the pelvic sidewalls via the lymphatic and capillary systems, which would allow for the anesthetic agent to come in direct contact with the nerve plexuses that innervate the pelvic structures. Safety of the technique has been proven over the years, given that it is widely used during office procedures that involve manipulation of the cervix. Although much of the focus regarding reducing postoperative pain has been centered on the abdominal wall and port sites, it is undeniable that a significant portion of pain actually arises from the pelvic surgical site; particularly since laparoscopic trocars have become smaller, resulting in less trauma. Our aim is to determine if infiltrating the cervical stroma with local anesthetic prior to performing a hysterectomy will reduce postoperative pain scores, and hence increase patient satisfaction.

Methods

Study design

This is a prospective randomized controlled trial in which patients that are scheduled to undergo a laparoscopic hysterectomy would be allocated to one of two groups: Paracervical block with local anesthetic (bupivacaine 0.5%), or placebo. This would be achieved using block randomization. The intervention would be performed after the patient is under general anesthesia, prior to starting the surgery. Patients would be consented in the office or preoperative area (before receiving sedatives). As far as the intervention itself, it would consist of injecting 10 mL of 0.5% bupivacaine into the cervical stroma at 3 and 9 o'clock, which is standard technique for para-cervical block. The remainder of the procedure will then continue in a regular fashion. Alternatively, patients in the control group will be injected with 10 mL of normal saline. The surgeon would be blinded as to patient allocation. The formulations (saline or bupivacaine) will be previously prepared in a syringe in the operating room by a member of the research time prior to beginning the procedure. At the end of the case, pain will be assessed using a visual analogue scale with a range from 0 to 10 (Wong-Baker faces - appendix 1) by one of the researches who will also be blinded to the group. This will be done at 30 and 60 minutes after surgical stop time. Additional pain control in the PACU will be standardized to all patients.

Study Subjects

Subjects will be selected based mainly on the fact they are undergoing a hysterectomy.

Sample Size

Investigators expect to detect a 25% reduction in pain reported on the visual analogue scale (VAS). Based on previous publications, it was determined that the mean VAS pain score after a laparoscopic hysterectomy is 5 with a standard deviation of 1.5. In order to detect the expected change after the proposed intervention, with a significance level of 5% and a power of 80%, a sample of 46 patients is required.

Data Collection

Data points to be collected are as follows:

* Age
* BMI
* Operating time
* History of cesarean deliveries
* Preoperative indication for surgery (pain, prolapse, tumor, bleeding, etc)
* Procedures performed (if ovaries/tubes were removed, if robotic assistance was used, if any additional procedures that are exceptions from the exclusion criteria were performed).
* Specimen weight
* Uterine pathology
* Pain score at 30 minutes (see appendix 1 for Wong-Baker scale)
* Pain score at 60 minutes
* Number of days in the hospital (zero if discharged on same-day)

Data Handling

A master key will be generated during randomization. It will contain patient initials and medical record number, and an individual code. Only the primary investigator will have access to this master key. A separate de-identified database using the individual code as index will be used for collection of all data points. The data that can be collected on the day of surgery (baseline characteristics, operating time, pain scores, etc) will be collected that day using a standardized form (appendix 2). This will later be transferred to the de-identified database. Using the master key, investigators will research pathology reports when available to complete final data points (uterine weight, histology, etc).

The data-collection sheets will be destroyed as soon as they are transferred into the de-identified database.

Data Analysis

Investigators will use T-Student tests to assure groups are homogenous to age, BMI, operating time, history of cesarean deliveries, and uterine weight. ChiSquare and Ancova analysis will be utilized to determine if there is a significant difference in reported pain scores between groups. Investigators will also stratify subjects based on uterine weight, history of cesarean delivery, additional procedures, etc. and determine if this has an effect on the reported pain scores.

Time Frame

Investigators expect to be able to consent and enroll at least two patients per week (average range of hysterectomy procedures per week from the surgeons that will participate is 5-10). Investigators expect the data collection phase to span over 30 weeks approximately.

Strength/Innovation

Patient satisfaction is a center point in today's healthcare. Faster recovery with less discomfort is not only standard of care, but may also translate into major economic advantages, such as less narcotic use and a decreased rate of postoperative admission. Using this technique as an adjuvant treatment for pain after laparoscopic hysterectomies has never been explored. There is data published for similar procedures, which demonstrates a clear benefit. If this study demonstrates significant improvement in pain scores, it has the potential to change standard of care for pain control during hysterectomy procedures.

Limitations

The main confounding factors are difference in operating style between surgeons and baseline surgical characteristics (large uteri that may require more dissection and tissue manipulation, etc.). To control for this investigators are only recruiting patients from 3 surgeons who have a similar operating technique. In addition to this, investigators are documenting operating time and specimen weight, which can be used to compare both groups and assure that they are homogeneous to these potential confounders. Further analysis will also be made specifically stratifying the data based on these characteristics.

Risks

The risks of the procedure are minimal. Regarding possible adverse reactions to the local anesthetic, there is no additional risk given that this is already routinely administered during surgery. Patients will be screened to confirm they do not have a history of allergies to the medication. Possible reactions include hypotension, bradycardia, headaches, tremors, etc. The paracervical block is routinely performed in the office setting before most invasive procedures involving the cervix, and risks are minimal, similar to those involving any subdermal injection. Possible risks include bleeding from injection site.

There is also the potential risk of accidental disclosure of the health information that will be collected.

Benefits

This study may find new methods of improving postoperative analgesia for patients undergoing minimally invasive hysterectomy procedures which may lead to less narcotic use, faster discharge from hospital, and greater satisfaction.

Costs

There is no additional costs. Local anesthetic and saline are products that are routinely used during all laparoscopic hysterectomy surgeries. The additional operating time it would take to perform the block is also negligible, since it is a procedure that can be accomplished in less than 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing laparoscopic hysterectomy with or without salpingoophorectomy for benign indications
* Undergoing laparoscopic hysterectomy with robotic assistance with or without salpingoophorectomy for benign indications
* Between 18 and 60 years of age

Exclusion Criteria:

* Intraoperative detection of malignancy
* Undergoing additional procedures at the time of surgery (except prophylactic McCall culdoplasty/uterosacral ligament suspension, excision of endometriosis, appendectomy, cystoscopy)
* Inability to perform paracervical block due to anatomic abnormalities (absent/flush cervix)
* Known allergy/sensitivity to bupivacaine
* Intraoperative bowel injury, bladder injury, ureter injury or major vessel injury that required repair.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Radtke, MD, Principal Investigator — UT College of Medicine MIGS Fellow & Faculty
Locations (1):
- Erlanger Medical Center, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Acton JN, Salfinger SG, Tan J, Cohen PA. Outcomes of Total Laparoscopic Hysterectomy Using a 5-mm Versus 10-mm Laparoscope: A Randomized Control Trial. J Minim Invasive Gynecol. 2016 Jan;23(1):101-6. doi: 10.1016/j.jmig.2015.09.001. Epub 2015 Sep 11. PMID 26371370
- [Background] Centini G, Calonaci A, Lazzeri L, Tosti C, Palomba C, Puzzutiello R, Luisi S, Petraglia F, Zupi E. Parenterally administered moderate sedation and paracervical block versus general anesthesia for hysteroscopic polypectomy: a pilot study comparing postoperative outcomes. J Minim Invasive Gynecol. 2015 Feb;22(2):193-8. doi: 10.1016/j.jmig.2014.09.008. Epub 2014 Nov 13. PMID 25265887
- [Background] Donnez O, Donnez J, Dolmans MM, Dethy A, Baeyens M, Mitchell J. Low Pain Score After Total Laparoscopic Hysterectomy and Same-Day Discharge Within Less Than 5 Hours: Results of a Prospective Observational Study. J Minim Invasive Gynecol. 2015 Nov-Dec;22(7):1293-9. doi: 10.1016/j.jmig.2015.06.021. Epub 2015 Jul 11. PMID 26169246
- [Background] Golembiewski J, Dasta J. Evolving Role of Local Anesthetics in Managing Postsurgical Analgesia. Clin Ther. 2015 Jun 1;37(6):1354-71. doi: 10.1016/j.clinthera.2015.03.017. Epub 2015 Apr 10. PMID 25866297
- [Background] Long JB, Eiland RJ, Hentz JG, Mergens PA, Magtibay PM, Kho RM, Magrina JF, Cornella JL. Randomized trial of preemptive local analgesia in vaginal surgery. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jan;20(1):5-10. doi: 10.1007/s00192-008-0716-6. Epub 2008 Oct 2. PMID 18830553
- [Background] Ng A, Swami A, Smith G, Davidson AC, Emembolu J. The analgesic effects of intraperitoneal and incisional bupivacaine with epinephrine after total abdominal hysterectomy. Anesth Analg. 2002 Jul;95(1):158-62, table of contents. doi: 10.1097/00000539-200207000-00028. PMID 12088961
- [Background] O'Neal MG, Beste T, Shackelford DP. Utility of preemptive local analgesia in vaginal hysterectomy. Am J Obstet Gynecol. 2003 Dec;189(6):1539-41; discussion 1541-2. doi: 10.1016/j.ajog.2003.10.691. PMID 14710057
- [Background] Penninx JP, Mol BW, Bongers MY. Endometrial ablation with paracervical block. J Reprod Med. 2009 Oct;54(10):617-20. PMID 20677480
- [Background] Skensved H. Combining Paracervical Block With a Complete Fundal Block Significantly Reduces Patients' Perception of Pain During Radio-Frequency Endometrial Ablation in an Office Setting. J Minim Invasive Gynecol. 2015 Nov-Dec;22(6S):S45. doi: 10.1016/j.jmig.2015.08.124. Epub 2015 Oct 15. No abstract available. PMID 27679246
- [Background] Tangsiriwatthana T, Sangkomkamhang US, Lumbiganon P, Laopaiboon M. Paracervical local anaesthesia for cervical dilatation and uterine intervention. Cochrane Database Syst Rev. 2013 Sep 30;2013(9):CD005056. doi: 10.1002/14651858.CD005056.pub3. PMID 24085642
- [Background] ACOG Committee Opinion No. 444: choosing the route of hysterectomy for benign disease. Obstet Gynecol. 2009 Nov;114(5):1156-1158. doi: 10.1097/AOG.0b013e3181c33c72. PMID 20168127
- [Background] Wong-Baker FACES Foundation (2016). Wong-Baker FACES® Pain Rating Scale. Retrieved 11/10/2016 with permission from http://www.WongBakerFACES.org
- [Background] Mercier RJ, Zerden ML. Intrauterine anesthesia for gynecologic procedures: a systematic review. Obstet Gynecol. 2012 Sep;120(3):669-77. doi: 10.1097/AOG.0b013e3182639ab5. PMID 22914480
- [Derived] Radtke S, Boren T, Depasquale S. Paracervical Block as a Strategy to Reduce Postoperative Pain after Laparoscopic Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2019 Sep-Oct;26(6):1164-1168. doi: 10.1016/j.jmig.2018.12.001. Epub 2018 Dec 6. PMID 30528725

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.50 (9.8) | 46 (10.4) | 46.24 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 41
BMI [Mean (Standard Deviation); unit: kg/m^2] | 35.05 (9.8) | 32.75 (9.8) | 33.87 (9.7)
history of csection [Count of Participants; unit: Participants] | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Pain Reported on the Visual Analogue Scale (VAS) at 30 Minutes Postoperative
Description: Scale used is the Visual analogue scale for pain. Scale ranges from 0 being no pain, to 10 being worse pain ever experienced.
Time Frame: 30 minutes post-operative stop time
Measure: Mean (Standard Deviation); unit: VAS scale 0-10
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 20 | 21
VAS scale 0-10 | 5.7 (2.8) | 3.2 (3.4)

2. Primary Outcome: Pain Reported on the Visual Analogue Scale (VAS) at 60 Minutes Postoperative
Description: Postoperative pain score on the Visual analgoue scale at 60 minutes from surgical stop time. Scale ranges from 0 being no pain, to 10 being worse pain ever experienced.
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: VAS scale 0-10
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 20 | 21
VAS scale 0-10 | 5.9 (3.0) | 2.3 (2.8)

ADVERSE EVENTS:
Time Frame: 30 days from enrollment
Description: Reaction to local anesthetic is the main adverse event expected. No adverse reactions were observed.
Arm/Group | Control Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT03027661/Prot_SAP_000.pdf